CLINICAL TRIAL: NCT04219800
Title: Reduced Occupational Sitting in Type 2 Diabetes Using mHealth (Mobile Health)
Acronym: ROSEBUD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Collaborators: Norrbottens County Council (Other Government); Vastra Gotaland Region (Other Government); Region Östergötland (Other); Region Stockholm (Other Government); Region Örebro County (Other); Region Västerbotten (Other Government); Region Jämtland Härjedalen (Other)
Responsible Party: Principal Investigator, Patrik Wennberg, Associate professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-05383
Record Dates: First submitted 2020-01-02; First posted 2020-01-07 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Experimental): 1. Activity tracker armband (Garmin Vivofit); warns of prolonged sitting and counts daily steps.
  2. SMS text messages; reminds of activity breaks.
  3. Mobile video instruction for standing pause gymnastics.
  Interventions: Behavioral: Patient-centered counselling and written material; Behavioral: mHealth
- Control (Other): Patient-centered counselling and written material regarding occupational sedentary behaviour, with telephone follow-ups after 1 and 5 weeks.
  Interventions: Behavioral: Patient-centered counselling and written material

INTERVENTIONS:
Behavioral: Patient-centered counselling and written material — Patient-centered counselling and written material regarding occupational sedentary behaviour, with telephone follow-ups after 1 and 5 weeks.
Behavioral: mHealth — 1. Activity tracker armband (Garmin Vivofit); warns of prolonged sitting and counts daily steps.
  2. SMS text messages; reminds of activity breaks.
  3. Mobile video instruction for standing pause gymnastics.
  Arms: mHealth

SUMMARY:
Type 2 diabetes mellitus (T2DM) patients are suboptimal treated due to low uptake of physical activity. Recent research shows promising beneficial health effects from reducing sitting time by regular short bouts of light-intensity physical activity. These findings open up for a new focus in T2DM treatment but conclusive evidence is missing as studies have been short-term trials, mainly conducted in laboratory environments. Recent research suggest that reduced sitting and increased physical activity can be supported at a low cost by mHealth (mobile health) technology such as activity tracker armbands that warns of prolonged sitting and SMS text messages that reminds of activity breaks.

The overarching purpose of the project is to evaluate the effects of an intervention aimed to reduce occupational sitting in T2DM using mHealth (mobile health). It is hypothesized that the intervention will lead to (1) Activity changes - reduced sitting time and/or increased number of steps (primary outcome measures) and (2) Health effects - lower fatigue, improved health-related quality of life, reduced cardiometabolic risk, less sick leave, less medication, less musculoskeletal problems (secondary outcome measures)

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Melltitus
* 40-64 years
* HbA1c 48-100 mmol/mol
* BMI ≥ 25 kg/m2
* Working at least 75% of full-time in a mainly seated job.

Exclusion Criteria:

* Pregnancy
* Regular vigorous intensity exercise
* Severe disease or for other reason unable to follow the study protocol

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sitting time | 12 months
  Assessed by activPAL3 thigh-worn accelerometer

SECONDARY OUTCOMES:
Steps | 12 months
  Assessed by activPAL3 thigh-worn accelerometer
Fatigue | 12 months
  MFI-20 questionnaire
Health-related quality of life | 12 months
  RAND-36 questionnaire
Cardiometabolic composite score (CCMR) | 12 months
  Will be determined by summing z-scores ([value-mean]/SD) of waist circumference (cm), mean arterial pressure (mmHg), HbA1c (mmol/mol), the inverse of HDL (mmol/L) and triglycerides (mmol/L), using sex-specific means and SDs
Sick leave | 12 months
  Assessed by diary
Medications | 12 months
  Total use of medications
Musculoskeletal problems | 12 months
  NRS questionnaire

OTHER OUTCOMES:
General self-efficacy | 12 months
  GSE-10 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Wennberg, Principal Investigator — Umeå University
Locations (6):
- Sweden (6):
  - Björkskatans Hälsocentral, Luleå, Norrbotten County
  - Hallsbergs hälsocentral, Hallsberg
  - Kärna Vårdcentral, Linköping
  - Clinical Research Centre, Östersund
  - Torsviks Vårdcentral, Stockholm
  - Clinical Research Centre, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Syrjala MB, Bennet L, Dempsey PC, Fharm E, Hellgren M, Jansson S, Nilsson S, Nordendahl M, Rolandsson O, Radholm K, Ugarph-Morawski A, Wandell P, Wennberg P. Health effects of reduced occupational sedentary behaviour in type 2 diabetes using a mobile health intervention: a study protocol for a 12-month randomized controlled trial-the ROSEBUD study. Trials. 2022 Jul 27;23(1):607. doi: 10.1186/s13063-022-06528-x. PMID 35897022